CLINICAL TRIAL: NCT03370432
Title: Associations Between Genetically Determined Low Vitamin D Level, Vitamin D Intake and Risk of Colorectal Cancer in a Prospective Case-cohort Study in Danes
Brief Title: Vitamin D, Genes and Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Vibeke Andersen, Clinical Professor, University of Southern Denmark
Other Study IDs: 19-Dvit
Record Dates: First submitted 2017-12-06; First posted 2017-12-12 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Colorectal Cancer
Keywords: Vitamin D; GC; CYP2R1; Gene-environment interaction; prospective case-cohort study; single nucleotide polymorphisms; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA extracted from buffy coeats
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Colorectal cancer cases: 1038 participants diagnosed with colorectal cancer from the Diet, Cancer and Health cohort.
  Interventions: Other: Observational
- Sub-cohort members: 1857 persons randomly selected within the full cohort at time of entry into the Diet, Cancer and Health cohort. These participants serve as controls for the colorectal cancer cases.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Information on diet, lifestyle, weight, height, medical treatment, environmental exposures, and other socio-economic factors were collected at enrolment using questionnaires and interviews

SUMMARY:
The aim of this study is to investigate the interaction between intake of vitamin D and polymorphisms in GC and CYP2R1 in relation to risk of colorectal cancer in a Danish prospective cohort study.

DETAILED DESCRIPTION:
The association between vitamin D and incidence of colorectal cancer (CRC) has been thoroughly investigated in both observational and experimental studies, but the results are conflicting. Genetic epidemiology is an advantageous alternative to randomized, clinical trials for ethical and economic reasons.

The aim of this study is to investigate whether polymorphisms in GC and CYP2R1 that predicts 25-hydroxycholecalciferol (25(OH)D) concentrations after both ultraviolet B radiation and consumption of vitamin D3-fortified bread and milk in Danes are associated with risk of CRC; and further, to examine whether intake of vitamin D through diet and supplementation alter the risk of CRC.

Data are retrieved from the Danish prospective "Diet, Cancer and Health" study encompassing 57,053 persons which were recruited between 1993 to 1997. Between 1994 and 31th December 2009, 1038 CRC cases has been diagnosed. A sub-cohort of 1857 persons has been randomly selected within the full cohort at time of entry into the cohort. The study design is a nested case-cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Born in Denmark
* No previous cancers at study entry
* Age between 50-64

Exclusion Criteria:

* Previous or present cancer(s) at study entry

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The Diet, Cancer and Health study is an ongoing Danish cohort study designed to investigate the relation between diet, lifestyle and cancer risk. The cohort consists of 57,053 persons, recruited between December 1993 and May 1997. All the subjects were born in Denmark, and the individuals were 50 to 64 years of age and had no previous cancers at study entry. Blood samples, anthropometric measures and questionnaire data on diet and lifestyle were collected at study entry.
  The present study uses a nested case-cohort design. Follow-up is based on population-based cancer registries. Between 1994 and 31th December 2009, 1038 CRC cases were diagnosed. A sub-cohort of 1857 persons has randomly been selected within the full cohort at time of entry into the cohort.
Sampling Method: Non-Probability Sample
Enrollment: 2895 (Actual)
Dates: Start 1993-12 (Actual); Primary Completion 1997-05 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Incidence of colorectal cancer in the DCH cohort | Between 1994 and 31th December 2009
  Risk of coloractal cancer compared to healthy sub-cohort members and interaction with Vitamin D metabolizing genes and vitamin D intake

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Andersen, MD, PhD, Study Director — University of Southern Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tjonneland A, Olsen A, Boll K, Stripp C, Christensen J, Engholm G, Overvad K. Study design, exposure variables, and socioeconomic determinants of participation in Diet, Cancer and Health: a population-based prospective cohort study of 57,053 men and women in Denmark. Scand J Public Health. 2007;35(4):432-41. doi: 10.1080/14034940601047986. PMID 17786808
- [Derived] Kopp TI, Vogel U, Andersen V. Associations between common polymorphisms in CYP2R1 and GC, Vitamin D intake and risk of colorectal cancer in a prospective case-cohort study in Danes. PLoS One. 2020 Feb 3;15(2):e0228635. doi: 10.1371/journal.pone.0228635. eCollection 2020. PMID 32012190
- See also: Description of the Diet, Cancer and Health cohort — https://www.cancer.dk/forskning/center-for-kraeftforskning/kost-gener-miljoe/kost-kraeft-helbred/